CLINICAL TRIAL: NCT03729310
Title: Comparison of Two Steroid Nasal Implants Following Endoscopic Sinus Surgery for Chronic Rhinosinusitis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1802018943
Record Dates: First submitted 2018-11-01; First posted 2018-11-02 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Chronic Sinusitis; Rhinosinusitis
Keywords: Propel Implant; Nasopore; Triamcinolone
MeSH Terms: conditions — Rhinosinusitis | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: Each subject will have both treatments (Propel and Nasopore), with one treatment on one side and the other treatment on the opposite side. The treatment for the right and left cavity will be selected in a randomized fashion (using opaque envelopes to assign each treatment to a respective ethmoid cavity).
Who Masked: Participant
Masking Description: Subjects will not have access to what treatment each cavity received through randomization. The information will be available should an emergency arise that would require the treating physician to know this information in order to best treat the subject. The subjects right to access this information will be reinstated when the study period is over (12 weeks after surgery).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Propel Implant (Other): The Propel 'implant' is composed of small, flexible tubes which dissolve while releasing Mometasone which is one type of steroid. This application has been approved for use by the FDA.
  Interventions: Device: Propel 'implant'
- Nasopore soaked with triamcinolone (Other): This "packing' is a sponge-like material which dissolves while releasing triamcinolone, which is another type of steroid. Triamcinolone has been approved for use topically elsewhere on the body, although the specific use of Triamcinolone in the sinuses has not been approved by the FDA.
  Interventions: Drug: Triamcinolone; Device: Nasopore

INTERVENTIONS:
Device: Propel 'implant' — The Propel 'implant' is composed of small, flexible tubes which dissolve while releasing Mometasone which is one type of steroid. This application has been approved for use by the FDA.
  Arms: Propel Implant
Drug: Triamcinolone — Triamcinolone has been approved for use topically elsewhere on the body, although the specific use of Triamcinolone in the sinuses has not been approved by the FDA.
  Arms: Nasopore soaked with triamcinolone
Device: Nasopore — This "packing' is a sponge-like material which dissolves while releasing triamcinolone.
  Arms: Nasopore soaked with triamcinolone

SUMMARY:
The purpose of this study is to learn whether there is a difference in postoperative (after surgery) endoscopic appearance of the sinus cavities (the way that the sinuses look through a camera) between sinuses that receive one of two types of resorbable steroid eluting sinus packing (a sponge-like material which dissolves within several days while releasing a steroid): 1) Propel Implant or 2) Nasopore soaked with triamcinolone at the time of endoscopic sinus surgery (ESS) for chronic rhinosinusitis.

DETAILED DESCRIPTION:
1. The Propel 'implant' is composed of small, flexible tubes which dissolve while releasing Mometasone which is one type of steroid. This application has been approved for use by the FDA.
2. Nasopore soaked with triamcinolone. This "packing' is a sponge-like material which dissolves while releasing triamcinolone, which is another type of steroid. Triamcinolone has been approved for use topically elsewhere on the body, although the specific use of Triamcinolone in the sinuses has not been approved by the FDA.

Both of these procedures are currently used regularly by Dr. Pearlman in practice at the conclusion of ESS for treatment of chronic rhinosinusitis. As standard of care, treatment is determined intraoperatively (during surgery), at the discretion of the surgeon. In this study, each subject will have both treatments (one in each cavity). The 'experimental' aspect relates to directly comparing the two procedures.

This research study is being done because there is currently a lack of consensus regarding the optimal nasal packing regimen. There have been no comparison studies and practice patterns vary widely. Our study looks to compare the Propel implant to Nasopore packing soaked in Triamcinolone.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients undergoing endoscopic sinus surgery for the treatment of chronic rhinosinusitis refractory to medical management

Exclusion Criteria:

* Patients ineligible for informed consent
* Patients unwilling or unable to comply with the postoperative visits necessary for data collection
* Patients with a history of intolerance to triamcinolone
* Patients with suspected systemic inflammatory disease, cystic fibrosis, and any contraindication to systemic corticosteroids.
* As standard of care, the PI does not operate on pregnant patients. A pregnant patient would not be a candidate for the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change from Pre-operative score in Patient's nasal endoscopy, as measured by Perioperative Sinus Endoscopy (POSE) Scores | Pre-operatively; Post-operatively at 1 week, 3 weeks, 6 weeks, 12 weeks.
  Validated endoscopy grading score.The score is calculated by determining several characteristics of the appearance of the sinus cavities. The score ranges from 0-32 (or 0-40 if frontal and sphenoid sinuses are opened at the time of surgery). A higher score indicates more severe disease.

SECONDARY OUTCOMES:
Change from Pre-operative score in Patient's nasal endoscopy, as measured by the Lund-Kennedy Endoscopic Score. | Pre-operatively; Post-operatively at 1 week, 3 weeks, 6 weeks, 12 weeks.
  The score is calculated by determining the amount of polyp, edema, and secretion in the nasal cavity on both sides. The score ranges from 0-12, with higher scores indicating more severe disease.
Change from Pre-operative score in Patient's sinonasal quality of life, as measured by SNOT-22 (Sino-nasal outcome test) | Pre-operatively; Post-operatively at 1 week, 3 weeks, 6 weeks, 12 weeks.
  Validated disease-specific quality of life questionnaire (22 questions). The score ranges from 0-110, with higher scores indicating more severe disease.

OTHER OUTCOMES:
Findings on the pre-operative CT scan, as measured by Lund-MacKay CT Scores | Pre-operatively
  The score is calculated by determining the amount of polyp, edema, and secretion in the nasal cavity on both sides. The score ranges from 0-12, with higher scores indicating more severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Pearlman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No